CLINICAL TRIAL: NCT07234695
Title: A Phase III, Randomized, Double-blinded Study of the Efficacy and Safety of LEvetiracetam to Prevent Seizures in Symptomatic Alzheimer's Disease in Adults With Down Syndrome (the LESS-AD Trial).
Brief Title: LEvetiracetam to Prevent Seizures in Symptomatic Alzheimer's Disease in Adults With Down Syndrome
Acronym: LESS-AD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); Hospital Universitario Marqués de Valdecilla (Other); Fundación CITA Alzheimer (Unknown); University Hospital Virgen de las Nieves (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IIBSP-LEV-2024-86; 2024-516148-24-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-02; First posted 2025-11-18 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Down Syndrome; Down Syndrome (DS); Down Syndrome (Trisomy 21); Alzheimer Dementia; Alzheimer Dementia (AD); Alzheimer Disease; Alzheimer Disease (AD); Alzheimer Blood Biomarkers; Epilepsy; Seizures
Keywords: Down syndrome; epilepsy; Alzheimer; dementia; levetiracetam; prevention; placebo-controlled; epileptic seizures; Alzheimer's disease markers; phase III; randomized; double-blind; bilateral tonic-clonic seizure; 217-pTau; NfL
MeSH Terms: conditions — Down Syndrome; Alzheimer Disease; Epilepsy; Seizures; Dementia; Epilepsy, Tonic-Clonic | interventions — Levetiracetam

STUDY DESIGN:
Intervention Model Description: This is a phase III, national, multicenter, randomized, double-blind, parallel-group, placebo-controlled clinical trial to evaluate the safety and efficacy of levetiracetam as a preventive treatment for epileptic seizures in adults with Alzheimer's disease associated with Down syndrome.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Clinical Research Associate, Project Manager, Data Manager
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levetiracetam 500 mg/12h (Experimental): Tablets for twice daily administration for 96 weeks. During the first 4 weeks of the treatment period, LEV, treatment will be administered 500mg/d (250mg/12h) to facilitate the compliance. During the last 4 weeks of the treatment period, LEV will be administered 500mg/d (250mg/12h) to enable a gradual withdrawal.
  Interventions: Drug: Levetiracetam 500mg
- Placebo (Placebo Comparator): Tablets for twice daily administration for 96 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levetiracetam 500mg — Use of Levetiracetam to prevent Seizures in Symptomatic Alzheimer's Disease in adults with Down syndrome (the LESS-AD trial)
  Arms: Levetiracetam 500 mg/12h
Drug: Placebo — Comparator
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether levetiracetam can prevent epileptic seizures in patients with Alzheimer's disease associated with Down syndrome. It will also analyze whether it can delay the neurodegeneration associated with this disease.

Patients will be randomly assigned to one of two groups: one group will receive the active drug (levetiracetam), and the other will receive a placebo.

Both groups will receive the treatment for 96 weeks. Each patient will participate for a total of 2 years and 5 months.

DETAILED DESCRIPTION:
This study is a clinical trial that will examine the efficacy and safety of a medication called levetiracetam in people with Down syndrome and Alzheimer's disease.

Adults with Down syndrome have a high risk of developing Alzheimer's disease. Epilepsy frequently coexists in these patients, and is associated with a worse clinical outcome. The early dysfunction of inhibitory interneuronal circuits, found in epilepsy, contributes to cognitive decline in Alzheimer's disease patients. Modifying this abnormal activity with levetiracetam could have potential benefits in the treatment of Alzheimer's disease, beyond its benefits on epileptic seizures' control and interictal epileptic activity recorded on EEG. Levetiracetam is a widely used drug with a proven safety profile, with more than 20 years of commercialization. This trial will evaluate the preventive benefit on the development of epileptic seizures in Alzheimer's disease associated with Down syndrome and, secondarily, its effect on cognitive decline and Alzheimer's disease markers. If the described benefits of levetiracetam use are independent of its antiepileptic effect, it could be a drug with a potential disease-modifying effect in Alzheimer's disease.

Primary objective:

To evaluate the efficacy of levetiracetam as a preventive measure for bilateral tonic-clonic seizures at 96 weeks in adults with Alzheimer's disease associated with Down syndrome.

Secondary objectives:

1. To quantify the time to the first bilateral tonic-clonic seizure between groups (levetiracetam vs. placebo).
2. To evaluate the incidence of mortality between groups (levetiracetam vs. placebo).
3. To study changes in biomarkers related to Alzheimer's disease:

   1. Functional changes (CAMDEX-DS)
   2. Cognitive changes (CAMCOG, mCRT)
   3. Plasma biomarkers (217-pTau, NfL)
   4. Brain structure (cortical thickness, hippocampal volume, gray matter volume)
   5. Epileptiform activity (EEG)
4. Safety: Incidence of adverse events and serious adverse events in the LEV vs. placebo groups.

A total of 120 participants will be included (60 per group).

The dose of levetiracetam to be used in this clinical trial is 1000 mg/day (two doses of 500mg each 12 hours) orally. During the first 4 weeks of the treatment period, LEV, treatment will be administered 500mg/d (250mg/12h) to facilitate the compliance. During the last 4 weeks of the treatment period, LEV will be administered 500mg/d (250mg/12h) to enable a gradual withdrawal.

Participants in placebo arm will receive placebo 1 capsule/12h during the 96 weeks of the treatment period.

The patients will have a total of 12 medical visits during their participation in the study. In those visits the following medical procedures will be carried out:

* Neuropsychological evaluation
* Blood analysis
* Magnetic resonance imaging (MRI)
* Electroencephalogram (EEG)

This study not only aims to improve the health and quality of life of people with Down syndrome but also to advance our general understanding of Alzheimer's disease, which could benefit more patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Down Syndrome (DS), either with a karyotype or a compatible typical phenotype.
* Age over 40 years at time of screening.
* Symptomatic Alzheimer's Disease (AD) dementia, based on change in functionality and neuropsychological tests' results. Different cut-off points will be established to diagnose dementia depending on the level of intellectual disability of the individual, according to previous experience (Benejam et al; 2020): in adults with mild intellectual disability, a CAMCOG-DS score of 80 and an mCRT score of 29 will be chosen, whereas values of 56 and 28, respectively, will be used in subjects with moderate intellectual disability. Doubtful cases (e.g., with compromised functionality, but without alteration in the neuropsychological assessment) or those unable to complete the evaluation will be categorized by consensus among expert clinicians, using all available clinical information.
* Willing and able caregiver who has daily contact with the study subject.
* Subjects and caregivers must be able to comply with the prescribed regimen of study treatment throughout the course of the study and meet a minimum required time commitment of biannual in-person visits.
* Any concurrent treatment for AD approved by the European Medicines Agency (EMA) must be stable for at least 30 days prior to screening and at least 60 days prior to study day 1. Other medications (except for those listed under exclusion criteria) are allowed as long as the dose is stable for 30 days prior to screening.
* Subjects and/or their caregivers must be able to provide their consent before participating in any study-related procedures.

Exclusion Criteria:

* Cognitive changes attributable to causes other than AD (for example, but not limited to, uncorrected visual or hearing deficit, severe, untreated sleep apnea or uncontrolled thyroid disorders).
* Previous history of adult-onset epileptic seizures (over 18 years old).
* Treatment with any kind of antiepileptic drugs, benzodiazepines, narcotics.
* Significant comorbidities or analytical abnormalities, such as:
* Any unstable and/or clinically significant medical condition likely to hamper the evaluation of safety and/or efficacy of the study (eg, moderate and/or severe untreated obstructive sleep apnea, clinically significant reduction in serum B12 or folate levels, clinically significant abnormalities of thyroid function, stroke, or other cerebrovascular conditions), as per investigator's judgement.
* Severe renal dysfunction (creatinine clearance < 30 mL/min), which would affect serum levetiracetam levels, or any other medical condition which is determined by the investigators to potentially create an undue risk for an adverse effect.
* Concomitant or past history psychiatric or neurologic disorder other than those considered to be related to AD (eg, head injury with loss of consciousness, symptomatic stroke, Parkinson's disease, severe carotid occlusive disease, transient ischemic attacks [TIAs]).
* Significant risk of suicide, defined using the C-SSRS as the subject answering "yes" to suicidal ideation questions 4 or 5 or answering "yes" to suicidal behavior within the past 12 months.
* Deviations from normal values for hematologic parameters, liver function tests, and other biochemical measures, judged to be clinically significant by the investigator.
* Participation in another clinical trial within 3 months of screening.
* Hypersensitivity to the active ingredient, other pyrrolidone derivatives, or any of the excipients
* Pregnant and breastfeeding patients

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Levetiracetam as a preventive treatment for epileptic seizures in adults with Alzheimer's disease associated with Down syndrome. | From enrollment to the end of treatment at 96 weeks
  Number (percentage) of subjects who do not develop a bilateral tonic-clonic epileptic seizure during the study treatment phase (96 weeks).

SECONDARY OUTCOMES:
Time to first bilateral tonic-clonic epileptic seizure | days
  Baseline (randomization) to first adjudicated epileptic seizure or censoring, up to 96 weeks.
All-cause mortality | percentage
  * All-cause mortality (number and percentage) - Time Frame: Baseline (randomization) to study completion, up to 96 weeks.
  * Alzheimer-related mortality (number and percentage) - Time Frame: Baseline (randomization) to study completion, up to 96 weeks.
Time to death | days
  Baseline (randomization) to death or censoring, up to 96 weeks.
Cognition | CAMCOG-DS: change from baseline and week 96.
  CAMCOG-DS (total score): change from baseline and week 96. Change from baseline visit in the CAMCOG-DS total score. Missing visits will be handled per the statistical analysis plan.
Plasma biomarkers -217p-tau | Change from baseline and week 96
  Plasma pTau-217-change (pg/mL) from baseline and week 96. Change from baseline in plasma pTau-217 concentration, quantified using the same laboratory and assay throughout the study.
Plasma biomarkers- NfL | At week 96
  Plasma Neurofilament light (NfL) (pg/mL) - Change from Baseline. Change from Baseline in plasma NfL concentration.
Neuroimaging GMV | At week 96
  Subcortical gray matter volume - change from Baseline (by region). Change from Baseline in volume (mm³) for 12 subcortical gray matter regions (left/right: amygdala, caudate, nucleus accumbens, pallidum, putamen, thalamus). Each region will be reported separately.
Neuroimaging- HV | Change at week 96
  Hippocampal volume (mm3)- Change from Baseline (left and right). Change from Baseline in hippocampal volume for the left and right hemispheres. Each hemisphere will be reported separately.
Neuroimaging- LVV | Week 96
  Lateral ventricle volume (mm3) - Change from Baseline (left and right). Change from Baseline in lateral ventricle volume for the left and right hemispheres. Each hemisphere will be reported separately.
Neuroimaging CTh | Week 96
  Cortical thickness (mm) - Change from Baseline (by region). Change from Baseline in cortical thickness (mm) for 34 left-hemispheric and 34 right-hemispheric cortical regions. Each region will be reported separately.
Electroencephalography (EEG) | At week 96.
  Presence of epileptiform/irritative graphoelements. Proportion of participants showing irritative graphoelements (spike-wave, polyspike-wave, sharp waves, focal or generalized slowing) per standardized EEG reading.
EEG- band power | At week 96
  EEG band power (µV²/Hz) - Change from Baseline. Change from Baseline in mean band power (δ, θ, α, β, γ) computed with a prespecified processing pipeline.
EEG sync | At week 96
  EEG synchronization/coherence (unitless index (0-1)) - Change from Baseline (by band). Change from Baseline in synchronization/coherence indices by frequency band (dimensionless 0-1) across predefined electrode pairs.
Safety of Levetiracetam | From enrollment to the end of treatment at 96 weeks
  The primary endpoints are number, type, frequency, and intensity of AEs evaluated until the end of treatment and assessment of tolerability during the medical visit, physical and neurological examination, vital signs, brain MRI assessment, suicidality (as measured with the C-SSRS), routine hematology and biochemistry evaluation in blood.
Incidence of adverse events (AEs) | At week 96
  Proportion (%) of participants:
  * with ≥1 treatment-emergent adverse events (TEAEs)
  * with TEAEs considered related to the treatment by the investigator
  * with ≥1 serious adverse events (SAEs) after first dose of treatment
  * who discontinue the study due to AEs
AEs- TEAE rate | Up to week 36
  TEAE rate- Rate of TEAEs per participant-year of exposure.
Maximum AE severity | At week 96
  Proportion of participants with at least one TEAE of maximum severity mild, moderate, or severe (% reported by category).
AEs- Dose interruptions | At week 96.
  Dose interruptions due to AEs. Proportion of participants with ≥1 levetiracetam dose interruption or reduction attributable to AEs.
Vital signs- BP | At week 96
  Systolic and diastolic blood pressure (mmHg)- Change from Baseline in systolic and diastolic blood pressure.
Vital signs- HR | At week 96
  Heart rate. Change from Baseline in resting heart rate (bpm).
Physical examination | Week 96
  Clinically significant abnormalities on physical/neurological exam. Proportion of participants with new or worsening clinically significant findings on physical or neurological examination.
Brain MRI safety | At week 96
  Clinically significant new MRI findings. Proportion of participants with new clinically significant MRI findings (e.g., edema, hemorrhage) vs Baseline.
Suicidality (C-SSRS) | Week 96
  Suicidal ideation or behavior (C-SSRS). Proportion of participants with any positive suicidal ideation or behavior signal on the C-SSRS.
Laboratory safety | At week 96
  Treatment-emergent hematology and biochemistry abnormalities:
  * Proportion of participants with ≥1 treatment-emergent hematology abnormality meeting predefined thresholds (e.g., CTCAE grade ≥2).
  * Proportion of participants with ≥1 treatment-emergent biochemistry abnormality meeting predefined thresholds (e.g., CTCAE grade ≥2).

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital Virgen de las Nieves, Granada, Andalusia
  - Fundación CITA Alzheimer, Donostia / San Sebastian, Basque Country
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital La Princesa, Madrid

IPD SHARING:
Plan to Share IPD: Undecided